CLINICAL TRIAL: NCT04725175
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single and Multiple Doses of PIPE-307 and Food Effect in Normal Healthy Volunteers
Brief Title: Phase I Study Evaluating Safety and Tolerability of Escalating Single and Multiple Doses of of PIPE-307 and Food Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PIPE-307-101
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All roles are masked with the exception of the pharmacist/dose preparer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PIPE-307 (Experimental)
  Interventions: Drug: PIPE-307
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: PIPE-307 — Single and multiple ascending oral doses of PIPE-307 tablets
  Arms: PIPE-307
Drug: Placebo oral tablet — Single and multiple ascending oral doses of matching Placebo tablets
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind study of PIPE-307 or placebo in normal healthy subjects. The study will be conducted in three parts: Part 1 will be a Single Ascending Dose (SAD) study enrolling approximately 48 subjects for a total duration of 6 weeks. Part 2 will be a Multiple Ascending Dose (MAD) study enrolling approximately 24 subjects for a total duration of 7 weeks, and part 3 will be a selected SAD cohort in a fed state to evaluate the effect of food on the bioavailability of PIPE-307, enrolling approximately 8 subjects from a selected SAD cohort for a duration of 6 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind study of PIPE-307 or placebo given as single and multiple escalating doses in normal healthy subjects. The study will be conducted in three parts: Part 1 will be a Single Ascending Dose (SAD) study enrolling approximately 48 subjects for a total duration of 6 weeks. Part 2 will be a Multiple Ascending Dose (MAD) study enrolling approximately 24 subjects for a total duration of 7 weeks, and part 3 will be a selected SAD cohort in a fed state to evaluate the effect of food on the bioavailability of PIPE-307, enrolling approximately 8 subjects from a selected SAD cohort for a duration of 6 weeks. Safety will be assessed by periodic measurement of vital signs, physical examinations, electrocardiograms, blood laboratory analyses and occurrence of adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (inclusive) at time of signing informed consent.
* BMI is between 18.0 and 32.0 kg/m2
* Male or female subjects with reproductive potential agree to comply with protocol-approved double barrier contraceptive method 30 days prior to first dose and up to 90 days post last dose
* Medically healthy with no clinically significant or relevant abnormalities in medical history physical exam, vital signs, electrocardiogram (ECG), or laboratory evaluations (hematology, chemistry, and urinalysis) as assessed by the Investigator.

Exclusion Criteria:

* Has a current or recurrent diseases that could affect the investigational medicinal product or affect clinical or laboratory assessments
* Experienced a significant systemic illness, as judged by the Investigator, within 30 days of the first dose
* Has a history of a significant medical, including hepatic and/or renal disease as outlined in the protocol, or psychiatric disorder that may require treatment or make the participant unlikely to fully complete the study or increase risk to the participant.
* History of alcohol or other substance abuse within the 12 months prior to dosing at the discretion of the Investigator
* Routine alcohol consumption meeting or exceeding protocol limits
* History of prior malignancy (except adequately treated non-melanoma skin cancer, carcinoma I-situ of the uterine cervix, ductal carcinoma in situ (DCIS), or localized prostate cancer
* Donated or lost more than 400ml of blood within 56 days or plasma within 14 days prior to screening
* Received an investigational agent with the last 30 days prior to dosing or within 5 half-lives of the investigational agent
* Use of any prescription medication, over-the-counter medication, vitamin or supplement, herbal or homeopathic preparations with 7 days or 5 half-lives prior to study drug administration, as determined by the Investigator. Hormone replacement therapy and hormonal contraception is permissible throughout the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Safety: Treatment-Emergent Adverse Events (TEAE) | From baseline to 7 days post dosing for SAD cohorts and 21 days post dosing for MAD cohorts
  Number of participants with TEAEs

SECONDARY OUTCOMES:
Safety: Cardiac repolarization using Fridericia-corrected QT interval (QTcF) | From baseline to 14 days post dose for SAD cohorts and 21 days post last dose for MAD cohorts
  Change in mean QTcF
Pharmacokinetics (PK): Blood concentration levels of PIPE-307 | From baseline to 14 days post dose for SAD cohorts and 21 days post last dose for MAD cohorts
PK: Urine concentration levels of PIPE-307 | From baseline on day 1 through day 2 for SAD cohorts, and from baseline on day 1 though day 7 for the MAD cohorts
Exploratory: Impact of PIPE-307 on Cogstate | From baseline to day 2 for SAD cohorts and from baseline to day 7 for MAD cohorts
  Cogstate tests have been designed, developed and validated to both identify and measure cognitive impairment, and to track or monitor cognitive changes. The tasks use novel visual and verbal stimuli to ensure assessment is cultural-neutral and not limited by a participant's level of education.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — Chief Medical Officer, Pipeline Therapeutics, Inc.
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia